CLINICAL TRIAL: NCT00427232
Title: Selective and Non-Selective Endothelin-Receptor Blockade in Coronary Artey Disease
Brief Title: Endothelin-Receptor Blockade in Coronary Heart Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: EK 242/2002
Record Dates: First submitted 2007-01-25; First posted 2007-01-26 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Coronary Vessels; Endothelins; Vascular Resistance
Keywords: coronary heart disease; endothelins; coronary angiography; blood flow velocity; fractional flow reserve, myocardial
MeSH Terms: conditions — Coronary Disease | interventions — cyclo(Trp-Asp-Pro-Val-Leu); BQ 788

INTERVENTIONS:
Drug: BQ-123 and BQ-788

SUMMARY:
Endothelin is a hormon that causes acute and chronic narrowing of heart vessels. The purpose of this study is to assess whether suppression of this activity by using two types of receptor antagonists can reduce this effect and thus improve blood supply of the heart muscle.

DETAILED DESCRIPTION:
Endothelin (ET) is the most potent vasoconstrictor known and plays a major role in the development of coronary artery disease as well as in acute vasoconstriction. This effect is mainly mediated by the vascular ET-A receptor, whereas the ET-B receptor mediates vasodilation and cleavage of ET. Currently, there are both selective ET-A antagonists and non-selective ET-A and ET-B antagonists under investigation. The aim of the study is to test the effect of ET-receptor blockade on the vasoreagibility of epicardial and intramyocardial coronary arteries in patients undergoing cardiac catheterization. We randomly use the selective ET-A receptor BQ-123 (Group A) and the combination of BQ-123 and the ET-B receptor antagonist BQ-788 (Group B). The tested infusion will be applied selectively into the assessed coronary artery by a special infusion catheter. To evaluate the morphometric changes we use quantitative coronary angiography to measure the diameter of the coronary artery before and after intracoronary infusion of the tested substances. Furthermore we will use Pressure Wire to measure the hemodynamic conditions before and after infusion, thus evaluating the epicardial and the intramyocardial blood perfusion.

Comparison: Coronary artery diameter as measured by quantitative angiography (minimal lumen diameter) and parameters indicative of epicardial and intramyocardial blood flow as determined by Pressure Wire (fractional flow reserver, coronary flow reserve, intramyocardial resistance) before and after ET-antagonist infusion will be compared.

ELIGIBILITY:
Inclusion Criteria:

* coronary artey disease
* stable angina pectoris
* male and post-menopausal female patients
* age above 19 years
* able and willing to conform to the requirements of the study
* provided written informed consent

Exclusion Criteria:

* severe focal coronary stenosis
* visually calcified stenosis
* aorto-ostial lesion location and unprotected left main stenosis
* pre-menopausal female patients
* diabetes mellitus
* unstable angina pectoris and/or acute Q-wave myocardial infarctaion within the past 72 hours
* current vasoactive medication
* previous percutaneous transluminal revascularization at the site of the target lesion
* lesion which has extremely angulated segments >90%
* vessel with escessive tortuosity of the proximal segment
* severe hypotension
* severely reduced left ventricular function
* severe carotid stenosis
* patients with pace maker
* patients with elevated liver enzymes
* patients simultaneously participating in another device or drug study
* inability of unwillingness to comply with the study protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26
Dates: Start 2003-05; Study Completion 2006-08

PRIMARY OUTCOMES:
minimal lumen diameter measured directly after infusion of the ET-antagonist(s)

SECONDARY OUTCOMES:
fractional flow reserve, coronary flow reserve, intramyocardial resistance measured directly after infusion of the ET-antagonist(s)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Neunteufl, MD, Principal Investigator — Dept. of Internal Medicine II, Medical University of Vienna
Locations (1):
- Dept. of Internal Medicine II, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Wexberg P, Sperker W, Morgenthaler NG, Heinzl H, Adlbrecht C, Plass C, Glogar HD, Lang IM, Neunteufl T. Inhomogeneous vasomotor effects of moderate selective and non-selective endothelin-receptor blockade in stable coronary artery disease. Heart. 2009 Aug;95(15):1258-64. doi: 10.1136/hrt.2008.158550. Epub 2009 May 3. PMID 19414437